CLINICAL TRIAL: NCT03343184
Title: Clinical Evaluation of Restorations With Filtek Bulk Fill, Associated With Single Bond Universal, With Different Adhesive Strategies
Brief Title: Clinical Evaluation of Bulk Fill Composite Restorations Associated to Universal Adhesive System
Acronym: FBFSBU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFFNFBULKANDUNIVERSAL2017
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: dentin bonding agents; tooth sensitivity; composite resin restoration
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SEE and incremental restoration (Active Comparator): 50 teeth will receive restorations using SEE Strategy and Incremental Restoration
  Interventions: Procedure: SEE Strategy and Incremental Restoration
- SEE and bulk restoration (Experimental): 50 teeth will receive restorations using SEE Strategy and Bulk Fill Restoration
  Interventions: Procedure: SEE Strategy and Bulk Fill Restoration
- SET and incremental restoration (Experimental): 50 teeth will receive restorations using SET Strategy and Incremental Restoration
  Interventions: Procedure: SET Strategy and Incremental Restoration
- SET and bulk restoration (Experimental): 50 teeth will receive restorations using SET Strategy and Bulk Fill Restoration
  Interventions: Procedure: SET Strategy and Bulk Fill Restoration

INTERVENTIONS:
Procedure: SEE Strategy and Incremental Restoration — 37% phosphoric acid will be applied during 30 seconds, only in enamel in 50 teeth. This acid will be removed using water, the cavity will be air-dried, and then, the adhesive will be brushed during 20 seconds in the cavity, will be air-dried during 5 seconds, and photoactivated during 10 seconds with Light Emission Diode (LED) light. Then, the Filtek Z350XT composite will be used in increments of no more than 2 mm, using the incremental restoration technique, and each increment will be photoactivated for 40 seconds.
  Arms: SEE and incremental restoration
Procedure: SEE Strategy and Bulk Fill Restoration — 37% phosphoric acid will be applied during 30 seconds, only in enamel in 50 teeth. This acid will be removed using water, the cavity will be air-dried, and then, the adhesive will be brushed during 20 seconds in the cavity, will be air-dried during 5 seconds, and photoactivated during 10 seconds with Light Emission Diode (LED) light. Then, the Filtek Bulk Fill composite will be used in increments of 4 mm, using the bulk restoration technique, and photoactivated for 40 seconds.
  Arms: SEE and bulk restoration
Procedure: SET Strategy and Incremental Restoration — no conditioning, the adhesive system will be used in 50 teeth, according to the manufacturer's instructions, in the self-etching mode. The adhesive system will be brushed during 20 seconds in the cavity, will be air-dried during 5 seconds, and photoactivated during 10 seconds with Light Emission Diode (LED) light. Then, the Filtek Z350XT composite will be used in increments of no more than 2 mm, using the incremental restoration technique, and each increment will be photoactivated for 40 seconds.
  Arms: SET and incremental restoration
Procedure: SET Strategy and Bulk Fill Restoration — no conditioning, the adhesive system will be used in 50 teeth, according to the manufacturer's instructions, in the self-etching mode. The adhesive system will be brushed during 20 seconds in the cavity, will be air-dried during 5 seconds, and photoactivated during 10 seconds with Light Emission Diode (LED) light. Then, the Filtek Bulk Fill composite will be used in increments of 4 mm, using the bulk restoration technique, and photoactivated for 40 seconds.
  Arms: SET and bulk restoration

SUMMARY:
Treatment clinical trial, randomized, controled, parallel, double-blinded, with four groups, that aims to evaluate the best application strategy when using a Universal Adhesive system, Single Bond Universal (3M ESPE, USA), in self-etch application mode, with or without enamel etching, associated wity a Bulk Fill Composite (Filtek Bulk Fill, 3M ESPE, USA), or with a conventional nanofilled composite (Filtek Z350 XT, 3M ESPE). Volunteers will be selected and recruited,following inclusion criteria and pre-established exclusion. All volunteers will be informed and sign a term of clarification and consent. 50 enrolled patients will receive 200 Class I or Class II dental restorations, made in four different ways, one from each experimental group, using the same universal self-etching adhesive system, with two application strategies, under the restorations that will use two different composites, a bulk fill composite, used in the bulk strategy, or a nanofilled composite, used in the traditional incremental strategy. Occlusal or Proximo-occlusal lesions will receive the selected adhesive system in 2 different protocols separated by groups. Group Self Etching and Bulk Fill (SETB), Group Selective enamel etching and Bulk Fill (SEEB), Group Self Etching and Filtek Z350XT (SETI), and Group Selective enamel etching and Filtek Z350XT (SEEI).Total time used in the restorations will be evaluated during the restorations. Immediate post-operative tooth sensitivity will be evaluated after one week. Restorations will be evaluated every 6 months for pain assessment, shape, fractures, staining or recurrent caries, using scores. To determine in which group each tooth will be enrolled, the authors will randomize the teeth.

DETAILED DESCRIPTION:
This is a Treatment clinical trial, randomized, controlled, parallel, double-blinded, with four groups, that aims to evaluate the best application strategy when using a Universal Adhesive system, Single Bond Universal (3M ESPE, USA), in self-etch application mode, with or without enamel etching, associated wity a Bulk Fill Composite (Filtek Bulk Fill, 3M ESPE, USA), or with a conventional nanofilled composite (Filtek Z350 XT, 3M ESPE). Volunteers will be selected and recruited, following inclusion criteria and pre-established exclusion. All volunteers will be informed and sign a term of clarification and consent. All 50 enrolled patients will receive 200 Class I or Class II dental restorations, made in four different ways, one from each experimental group, using the same universal self-etching adhesive system, with two application strategies, under the restorations that will use two different composites, a bulk fill composite, used in the bulk strategy, or a nanofilled composite, used in the traditional incremental strategy. All patients must have at only 20 teeth in function, must have at only 4 carious lesion in occlusal or proximo-occlusal face in posterior teeth or old restorations in the same faces, with problems, that need to be changed. Those lesions must be more than 2 mm deep, should have exposed dentin, and must have at only 50% of margins in enamel. Teeth should not present periodontal mobility. Firstly, the patient will be anesthetized locally with 3% Mepivacaine solution, followed by prophylaxis with pumice powder and water. All cavities will be washed and dried after these procedures for optimal selection of color, using a color scale. Then, the rubber dam isolation of the teeth to be restored will be held. Occlusal or Proximo-occlusal lesions will receive the selected adhesive system in 2 different protocols separated by groups. Group Self Etching and Bulk Fill (SETB): no conditioning, the adhesive system will be used in 50 teeth, according to the manufacturer's instructions, in the self-etching mode. The adhesive system will be brushed during 20 seconds in the cavity, will be air-dried during 5 seconds, and photoactivated during 10 seconds with Light Emission Diode (LED) light. Then, the Filtek Bulk Fill composite will be used in increments of 4 mm, using the bulk restoration technique, and photoactivated for 40 seconds; Group Selective enamel etching and Bulk Fill (SEEB): 37% phosphoric acid will be applied during 30 seconds, only in enamel in 50 teeth. This acid will be removed using water, the cavity will be air-dried, and then, the adhesive will be applied according to the manufacturer's instructions, as described in group SETB. Restorations will also be made as described in group SETB; Group Self Etching and Filtek Z350XT (SETI): no conditioning, the adhesive system will be used in 50 teeth, according to the manufacturer's instructions, in the self-etching mode. The adhesive system will be brushed during 20 seconds in the cavity, will be air-dried during 5 seconds, and photoactivated during 10 seconds with Light Emission Diode (LED) light. Then, the Filtek Z350XT composite will be used in increments of no more than 2 mm, using the incremental restoration technique, and each increment will be photoactivated for 40 seconds.; Group Selective enamel etching and Filtek Z350XT (SEEI): 37% phosphoric acid will be applied during 30 seconds, only in enamel in 50 teeth. This acid will be removed using water, the cavity will be air-dried, and then, the adhesive will be applied according to the manufacturer's instructions, as described in group SETI. Restorations will also be made as described in group SETI. Total time used in the restorations will be evaluated during the restorations. Immediate post-operative tooth sensitivity will be evaluated after one week. Restorations will be evaluated every 6 months for pain assessment, shape, fractures, staining or recurrent caries, using scores. To determine in which group each tooth will be enrolled, the authors will randomize the teeth.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have at only 20 teeth in function, must have at only 4 carious occlusal or proximo-occlusal lesions, or old restorations that need to be changed, in different teeth. Those lesions must be more than 2 mm deep, should have exposed dentin, and must have at only 50% of margins in enamel. Teeth should not present periodontal mobility.

Exclusion Criteria:

* Volunteers with periodontal disease; with gingival bleeding; use of anti-inflammatory drugs in the last 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Restoration Loss | Five years
  It will be evaluated the increase in the number of losses of dental restorations in the period of five years, verified by periodic visual clinical examination (6/6 months) based on the statement of difference of at least 25% in the amount of remaining restorations in the different groups.

SECONDARY OUTCOMES:
Marginal Pigmentation | Five years
  It will be evaluated the increase in the number of dental restorations with marginal pigmentation in the period of five years, verified by periodic clinical visual examination (6/6 months) based on the statement of difference of at least 25% in the amount of stained restorations in the different groups.
Post-Operative Hypersensitivity | Five years
  It will be evaluated the increase in the number of dental restorations with dentin hypersensitivity in the period of five years, verified by periodic clinical examination (6/6 months) based on the statement of difference of at least 25% in the amount of restorations with dentin hypersensitivity in the different groups.
Secondary Caries | Five years
  It will be evaluated the increase in the number of dental restorations with secondary caries in the period of five years, verified by periodic radiographic examination (6/6 months) based on the statement of difference of at least 25% in the amount of restorations with secondary caries in the different groups.

CONTACTS AND LOCATIONS:
Overall Officials: MARCOS O BARCELEIRO, DDS, PhD, Study Director — Universidade Federal Fluminense
Locations (1):
- Universidade Federal Fluminense - School of Dentistry, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pashley DH, Tay FR. Aggressiveness of contemporary self-etching adhesives. Part II: etching effects on unground enamel. Dent Mater. 2001 Sep;17(5):430-44. doi: 10.1016/s0109-5641(00)00104-4. PMID 11445211
- [Background] Perdigao J, Kose C, Mena-Serrano AP, De Paula EA, Tay LY, Reis A, Loguercio AD. A new universal simplified adhesive: 18-month clinical evaluation. Oper Dent. 2014 Mar-Apr;39(2):113-27. doi: 10.2341/13-045-C. Epub 2013 Jun 26. PMID 23802645
- [Background] Erhardt MC, Cavalcante LM, Pimenta LA. Influence of phosphoric acid pretreatment on self-etching bond strengths. J Esthet Restor Dent. 2004;16(1):33-40; discussion 41. doi: 10.1111/j.1708-8240.2004.tb00448.x. PMID 15259541
- [Background] Erickson RL, Barkmeier WW, Latta MA. The role of etching in bonding to enamel: a comparison of self-etching and etch-and-rinse adhesive systems. Dent Mater. 2009 Nov;25(11):1459-67. doi: 10.1016/j.dental.2009.07.002. Epub 2009 Aug 7. PMID 19665220
- [Background] Torii Y, Itou K, Nishitani Y, Ishikawa K, Suzuki K. Effect of phosphoric acid etching prior to self-etching primer application on adhesion of resin composite to enamel and dentin. Am J Dent. 2002 Oct;15(5):305-8. PMID 12537339
- [Background] Van Landuyt KL, Peumans M, De Munck J, Lambrechts P, Van Meerbeek B. Extension of a one-step self-etch adhesive into a multi-step adhesive. Dent Mater. 2006 Jun;22(6):533-44. doi: 10.1016/j.dental.2005.05.010. Epub 2005 Nov 21. PMID 16300826
- [Background] Abbas G, Fleming GJ, Harrington E, Shortall AC, Burke FJ. Cuspal movement and microleakage in premolar teeth restored with a packable composite cured in bulk or in increments. J Dent. 2003 Aug;31(6):437-44. doi: 10.1016/s0300-5712(02)00121-5. PMID 12878027
- [Background] Moorthy A, Hogg CH, Dowling AH, Grufferty BF, Benetti AR, Fleming GJ. Cuspal deflection and microleakage in premolar teeth restored with bulk-fill flowable resin-based composite base materials. J Dent. 2012 Jun;40(6):500-5. doi: 10.1016/j.jdent.2012.02.015. Epub 2012 Mar 3. PMID 22390980
- [Background] Roggendorf MJ, Kramer N, Appelt A, Naumann M, Frankenberger R. Marginal quality of flowable 4-mm base vs. conventionally layered resin composite. J Dent. 2011 Oct;39(10):643-7. doi: 10.1016/j.jdent.2011.07.004. Epub 2011 Jul 27. PMID 21801799
- [Background] van Dijken JW, Pallesen U. Randomized 3-year clinical evaluation of Class I and II posterior resin restorations placed with a bulk-fill resin composite and a one-step self-etching adhesive. J Adhes Dent. 2015 Feb;17(1):81-8. doi: 10.3290/j.jad.a33502. PMID 25625133
- [Background] Bayraktar Y, Ercan E, Hamidi MM, Colak H. One-year clinical evaluation of different types of bulk-fill composites. J Investig Clin Dent. 2017 May;8(2). doi: 10.1111/jicd.12210. Epub 2016 Jan 22. PMID 26800647
- [Background] van Dijken JW, Pallesen U. A randomized controlled three year evaluation of "bulk-filled" posterior resin restorations based on stress decreasing resin technology. Dent Mater. 2014 Sep;30(9):e245-51. doi: 10.1016/j.dental.2014.05.028. Epub 2014 Jun 21. PMID 24958689
- [Background] Swift EJ Jr, Perdigao J, Heymann HO, Wilder AD Jr, Bayne SC, May KN Jr, Sturdevant JR, Roberson TM. Eighteen-month clinical evaluation of a filled and unfilled dentin adhesive. J Dent. 2001 Jan;29(1):1-6. doi: 10.1016/s0300-5712(00)00050-6. PMID 11137632
- [Background] Cvar JF, Ryge G. Reprint of criteria for the clinical evaluation of dental restorative materials. 1971. Clin Oral Investig. 2005 Dec;9(4):215-32. doi: 10.1007/s00784-005-0018-z. No abstract available. PMID 16315023
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Clin Oral Investig. 2007 Mar;11(1):5-33. doi: 10.1007/s00784-006-0095-7. Epub 2007 Jan 30. PMID 17262225
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Dalton Bittencourt D, Ezecelevski IG, Reis A, Van Dijken JW, Loguercio AD. An 18-months' evaluation of self-etch and etch & rinse adhesive in non-carious cervical lesions. Acta Odontol Scand. 2005 Jun;63(3):173-8. doi: 10.1080/00016350510019874. PMID 16191912